CLINICAL TRIAL: NCT00951496
Title: A Phase III Clinical Trial of Bevacizumab With IV Versus IP Chemotherapy in Ovarian, Fallopian Tube and Primary Peritoneal Carcinoma
Brief Title: Bevacizumab and Intravenous or Intraperitoneal Chemotherapy in Treating Patients With Stage II-III Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01956; NCI-2011-01956 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 09-0724; CDR0000650601; GOG-0252 (Other: NRG Oncology); GOG-0252 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2009-08-01; First posted 2009-08-04 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-03

CONDITIONS: Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Fallopian Tube Undifferentiated Carcinoma; Malignant Ovarian Brenner Tumor; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Adenocarcinoma; Ovarian Transitional Cell Carcinoma; Ovarian Undifferentiated Carcinoma; Primary Peritoneal Clear Cell Adenocarcinoma; Primary Peritoneal Endometrioid Adenocarcinoma; Primary Peritoneal Serous Adenocarcinoma; Primary Peritoneal Transitional Cell Carcinoma; Primary Peritoneal Undifferentiated Carcinoma; Stage II Fallopian Tube Cancer AJCC v6 and v7; Stage II Ovarian Cancer AJCC v6 and v7; Stage IIA Fallopian Tube Cancer AJCC v6 and v7; Stage IIA Ovarian Cancer AJCC V6 and v7; Stage IIB Fallopian Tube Cancer AJCC v6 and v7; Stage IIB Ovarian Cancer AJCC v6 and v7; Stage IIC Fallopian Tube Cancer AJCC v6 and v7; Stage IIC Ovarian Cancer AJCC v6 and v7; Stage III Ovarian Cancer AJCC v6 and v7; Stage III Primary Peritoneal Cancer AJCC v7; Stage IIIA Ovarian Cancer AJCC v6 and v7; Stage IIIA Primary Peritoneal Cancer AJCC v7; Stage IIIB Ovarian Cancer AJCC v6 and v7; Stage IIIB Primary Peritoneal Cancer AJCC v7; Stage IIIC Ovarian Cancer AJCC v6 and v7; Stage IIIC Primary Peritoneal Cancer AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: conditions — Brenner Tumor | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (paclitaxel, carboplatin, bevacizumab) (Experimental): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and carboplatin IV over 30 minutes on day 1. Patients also receive bevacizumab IV over 30-90 minutes on day 1 in courses 2-6. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive bevacizumab alone in courses 7-22 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment
- Arm II (paclitaxel, bevacizumab, carboplatin IP) (Experimental): Patients receive paclitaxel as in Arm I and carboplatin IP on day 1. Patients also receive bevacizumab as in Arm I. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive bevacizumab alone as in Arm I.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment
- Arm III (paclitaxel IP, bevacizumab, cisplatin IP) (Experimental): Patients receive paclitaxel IV over 3 hours on day 1, cisplatin IP on day 2, and paclitaxel IP on day 8. Patients also receive bevacizumab as in Arm I. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive bevacizumab alone as in Arm I.
  Interventions: Biological: Bevacizumab; Drug: Cisplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; Zirabev
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm I (paclitaxel, carboplatin, bevacizumab)
Drug: Carboplatin — Given IP
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm II (paclitaxel, bevacizumab, carboplatin IP)
Drug: Cisplatin — Given IP
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm III (paclitaxel IP, bevacizumab, cisplatin IP)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Paclitaxel — Given IP
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm III (paclitaxel IP, bevacizumab, cisplatin IP)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies bevacizumab and intravenous (given into a vein) chemotherapy to see how well they work compared with bevacizumab and intraperitoneal (given into the abdominal cavity) chemotherapy in treating patients with stage II-III ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer. Monoclonal antibodies, such as bevacizumab, can block the ability of tumor cells to grow and spread by blocking the growth of new blood vessels necessary for tumor growth. Drugs used in chemotherapy, such as paclitaxel, carboplatin, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving bevacizumab together with intravenous chemotherapy is more effective than giving bevacizumab together with intraperitoneal chemotherapy in treating patients with ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if one or both of the proposed intraperitoneal chemotherapy regimens improves the progression-free survival (PFS) event rate compared to standard intravenous chemotherapy for first-line treatment of patients diagnosed with advanced stage ovarian, peritoneal or fallopian tube cancer.

II. If both intraperitoneal (IP) regimens significantly improve the PFS event rate compared to the standard regimen, then a second study objective is to determine whether IP cisplatin and intravenous (IV) paclitaxel on day one plus IP paclitaxel on day eight improves the PFS event rate when compared to the IP carboplatin and IV paclitaxel.

SECONDARY OBJECTIVES:

I. To determine if intraperitoneal chemotherapy reduces the overall death rate compared to standard intravenous chemotherapy.

II. To assess the frequency and severity of adverse events as defined by Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.

III. To compare the patient-reported outcomes on: Quality of Life (Function Assessment of Cancer Therapy-Ovarian-Trial Outcome Index [FACT-O-TOI]), Neuropathy (FACT-Gynecologic Oncology Group/Neurotoxicity [GOG/NTX4] scale), Abdominal discomfort (FACT-GOG/AD scale), Fatigue (FACIT-Fatigue scale), and Nausea (item from FACT-O-TOI).

IV. To assess the frequency and the reasons for early discontinuation of the study treatments.

TERTIARY OBJECTIVES:

I. To bank deoxyribonucleic acid (DNA) from whole blood for research and examine the association between single nucleotide polymorphisms (SNPs) and measures of clinical outcome including overall survival, progression-free survival and adverse events.

II. To bank archival tumor for research and examine the association between tumor markers and measures of clinical outcome including overall survival, progression-free survival and adverse events.

III. Patients will be encouraged to enroll on the companion translational research protocol (CEM0703 under development).

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and carboplatin IV over 30 minutes on day 1. Patients also receive bevacizumab IV over 30-90 minutes on day 1 in courses 2-6. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive bevacizumab alone in courses 7-22 in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive paclitaxel as in Arm I and carboplatin IP on day 1. Patients also receive bevacizumab as in Arm I. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive bevacizumab alone as in Arm I.

ARM III: Patients receive paclitaxel IV over 3 hours on day 1, cisplatin IP on day 2, and paclitaxel IP on day 8. Patients also receive bevacizumab as in Arm I. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive bevacizumab alone as in Arm I.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of epithelial ovarian, fallopian tube, or primary peritoneal carcinoma, stage II, III, or IV with either optimal (=< 1 cm residual disease) or suboptimal residual disease; in the event of a higher priority Phase III Gynecologic Oncology Group (GOG) protocol becoming available for suboptimal and/or stage IV patients, the eligibility of this study will narrow and exclude those patients at those participating institutions (11/02/2009)

  * Note: patients with suboptimal disease/and or stage IV will not be eligible as of April 1, 2011; they should be enrolled on GOG-0262 (03/14/11)
  * All patients must have a procedure for determining diagnosis of epithelial ovarian, fallopian tube, primary peritoneal, with appropriate tissue for histologic evaluation; the minimum surgery required is an abdominal surgery providing tissue for histologic evaluation and establishing and documenting the primary site and stage, as well as a maximal effort at tumor debulking; if additional surgery was performed, it should have been in accordance with appropriate surgery for ovarian or peritoneal carcinoma described in the GOG Surgical Procedures Manual (https://www.gog.fccc.edu/manuals/pdf/surgman.pdf) (11/02/2009)(08/16/2010)
* Patients with the following histologic epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma not otherwise specified (N.O.S.); however, the histologic features of the tumor must be compatible with a primary Müllerian epithelial adenocarcinoma; if doubt exists, it is recommended that the investigator should have the slides reviewed by an independent pathologist prior to entry; patients may have co-existing endometrial cancer so long as the primary origin of invasive tumor is ovarian or peritoneal; Note: patients with mucinous, low grade and clear cell disease are eligible unless there is a higher priority GOG trial open (11/02/2009) (08/16/2010)
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl, equivalent to Common Terminology Criteria for Adverse Events v3.0 (CTCAE) grade 1; this ANC cannot have been induced or supported by granulocyte colony stimulating factors
* Platelets greater than or equal to 100,000/mcl
* Creatinine no greater than institutional upper limits of normal (03/29/10)
* Bilirubin less than or equal to 1.5 x upper limit of normal (ULN) (CTCAE grade 1)
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) less than or equal to 2.5 x ULN (CTCAE grade 1)
* Alkaline phosphatase less than or equal to 2.5 x ULN (CTCAE grade 1)
* Neuropathy (sensory and motor) less than or equal to CTCAE grade 1
* Prothrombin time (PT) such that international normalized ratio (INR) is =< 1.5 x ULN (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a partial thromboplastin time (PTT) =< 1.5 times the upper limit of normal (heparin, Lovenox or alternative anticoagulants are acceptable); this corresponds to CTCAE version 3.0 grade 1 one or less (11/02/2009) (03/29/10)
* Patients with a GOG performance status of 0, 1, or 2
* Patients must be entered and treated within 12 weeks of their most recent surgery performed for the combined purpose of diagnosis, staging and/or cytoreduction; the first cycle of chemotherapy should not be given until at least seven days after the most recent major surgery, which allows 4 weeks to have elapsed prior to the first bevacizumab dose; (placement of venous or peritoneal access devices will be considered minor surgery) (03/29/10)
* Patients who have met the pre-entry requirements specified
* An approved informed consent and authorization permitting release of personal health information must be signed by the patient or guardian
* Patients in this trial may receive ovarian estrogen +/- progestin replacement therapy as indicated at the lowest effective dose(s) for control of menopausal symptoms at any time, but high dose progestin as an appetite stimulant should be avoided (03/29/10)

Exclusion Criteria:

* Patients with a current diagnosis of borderline epithelial ovarian tumor (formerly "tumors of low malignant potential") or recurrent invasive epithelial ovarian cancer treated with surgery only (such as those with stage IA or IB low grade lesions) are not eligible; patients with a prior diagnosis of a borderline tumor that was surgically resected and who subsequently develop an unrelated, new invasive epithelial ovarian or peritoneal primary cancer are eligible, provided that they have not received prior chemotherapy for any ovarian tumor
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies are excluded if there is any evidence of the other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy (11/02/2009)
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor including neo-adjuvant chemotherapy for their ovarian or primary peritoneal cancer are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients who have received any targeted therapy (including but not limited to vaccines, antibodies, tyrosine kinase inhibitors) or hormonal therapy for management of their epithelial ovarian or peritoneal primary cancer
* Patients with synchronous primary endometrial cancer, or a past history of primary endometrial cancer, are excluded, unless all of the following conditions are met: stage not greater than IB; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell or other FIGO grade 3 lesions
* Patients with acute hepatitis or active infection that requires parenteral antibiotics
* Patients with serious non-healing wound, ulcer, or bone fracture; this includes history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days; patients with granulating incisions healing by secondary intention with no evidence of fascial dehiscence or infection are eligible but require weekly wound examinations
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients with history or evidence upon physical examination of major central nervous system (CNS) disease (for example: primary brain tumor, metastatic cancer in the brain, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident [CVA, stroke], transient ischemic attack [TIA] or subarachnoid hemorrhage within six months of the first date of treatment on this study) (11/02/2009) (03/29/10)
* Patients with clinically significant cardiovascular disease; this includes:

  * Uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 90 mmHg
  * Myocardial infarction or unstable angina < 6 months prior to registration
  * New York Heart Association (NYHA) grade II or greater congestive heart failure
  * Serious cardiac arrhythmia requiring medication; this does not include asymptomatic atrial fibrillation with controlled ventricular rate, or past history of supraventricular tachycardia controlled with medications and that is asymptomatic (03/29/10)
  * CTCAE grade 2 or greater peripheral vascular disease (at least brief (< 24 hrs) episodes of ischemia managed non-surgically and without permanent deficit)
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies; patients with known allergy to Cremophor or polysorbate 80
* Patients with clinically significant proteinuria; urine protein should be screened by urine protein-creatinine ratio (UPCR); patients must have a UPCR < 1.0 to allow participation in the study
* Patients with or with anticipation of invasive procedures as defined below:

  * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to the first date of bevacizumab therapy (cycle 2)
  * Major surgical procedure anticipated during the course of the study; this includes, but is not limited to abdominal surgery (laparotomy or laparoscopy) prior to disease progression, such as colostomy or enterostomy reversal, interval or secondary cytoreductive surgery, or second look surgery
  * Core biopsy, within 7 days prior to the first date of bevacizumab therapy (cycle 2)
* Patients with GOG performance grade of 3 or 4
* Patients who are pregnant or nursing; patients of childbearing potential must agree to use contraceptive measures during study therapy and for at least six months after completion of bevacizumab therapy
* Patients who have received prior therapy with any anti-vascular endothelial growth factor (VEGF) drug, including bevacizumab
* Patients with clinical symptoms or signs of gastrointestinal obstruction and/ or those who require parenteral hydration and/or nutrition; patients with history or current diagnosis of inflammatory bowel disease are not eligible (12/20/10)
* Patients with medical history or conditions not otherwise previously specified which in the opinion of the investigator should exclude participation in this study; examples of this would be: persistent gastrointestinal symptoms resulting from clostridia difficile enterocolitis or bowel surgery which may increase gastrointestinal toxicity from bevacizumab; or hearing loss or neuropathy which would prevent tolerance to cisplatin, and paclitaxel administration; the investigator should feel free to consult the Study Chair or Study Co-Chairs for uncertainty in this regard (12/20/10)
* Patients with metastatic tumor in the parenchyma of the liver or lungs with proximity to large vessels which could make the patient as high risk of lethal hemorrhage during treatment with bevacizumab (i.e. hemoptysis, liver rupture) (11/02/2009)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1560 (Actual)
Dates: Start 2009-08-11 (Actual); Primary Completion 2016-01-11 (Actual); Study Completion 2016-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan L Walker, Principal Investigator — NRG Oncology
Locations (503):
- United States (503):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Marin General Hospital, Greenbrae, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Colorado Gynecologic Oncology Group, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - University of Colorado, Denver, Colorado
  - Rocky Mountain Gynecologic Oncology PC, Englewood, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Saint Vincent's Medical Center, Jacksonville, Florida
  - Southeast Gynecologic Oncology Associates, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - The Watson Clinic, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Bayfront Outpatient Health Clinic, St. Petersburg, Florida
  - Women's Cancer Associates, St. Petersburg, Florida
  - Northside Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Kootenai Cancer Center, Post Falls, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Cottage, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Associates in Oncology Hematology PC -Kensington, Kensington, Maryland
  - Maryland Oncology Hematology PA-Aquilino Cancer Center, Rockville, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Commonwealth Hematology Oncology PC-Worcester, Worcester, Massachusetts
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Luke's Hospital, Chesterfield, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - The Women's Oncology Center, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Island Gynecologic Oncology, Brightwaters, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Hospital Medical Center of Queens, Fresh Meadows, New York
  - Queens Hospital Center, Jamaica, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - NYU Winthrop Hospital, Mineola, New York
  - Mount Kisco Medical Group, Mount Kisco, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - University of Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Northern Virginia Pelvic Surgery Associates, Annandale, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - PeaceHealth Medical Group PC, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Cancer Institutes of Washington PLLC, Yakima, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Walker JL, Brady MF, Wenzel L, Fleming GF, Huang HQ, DiSilvestro PA, Fujiwara K, Alberts DS, Zheng W, Tewari KS, Cohn DE, Powell MA, Van Le L, Davidson SA, Gray HJ, Rose PG, Aghajanian C, Myers T, Alvarez Secord A, Rubin SC, Mannel RS. Randomized Trial of Intravenous Versus Intraperitoneal Chemotherapy Plus Bevacizumab in Advanced Ovarian Carcinoma: An NRG Oncology/Gynecologic Oncology Group Study. J Clin Oncol. 2019 Jun 1;37(16):1380-1390. doi: 10.1200/JCO.18.01568. Epub 2019 Apr 19. PMID 31002578

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was opened for accrual on July 27, 2009. Target accrual was about 1500 patients. The study was closed to enrollment on Nov 30, 2011 after enrolling 1560 individuals.
Pre-assignment Details: Eligibility was verified by a web-based procedure which reviewed all eligibility criteria prior to each subject's registration. Prior to treatment randomization patients were stratified by stage of disease and size of residual disease.
Groups:
- Arm I (Paclitaxel, Carboplatin, Bevcizumab IV): Six cycles of Paclitaxel 80mg/m2 IV over ' hours days 1, 8 and 15. Carboplatin AUC 6 IV on day 1, Bevacizumab 15mg/kg IV on day 1 beginning on cycle 2, followed by bevacizumab 15mg/kg for cycles 7-22.
- Arm II (Paclitaxel,carboplatinIP, Bevacizumab IP): Six cycles of Paclitaxel 80mg/m2 IV over 1 hour days 1, 8, and 15, Carboplatin AUC 6 IP on day1, Bevacizumab 15mg/kg IV on day 1 beginning on cycle 2 followed by bevacizumab 15mg/KG for cycles 7-22
- Arm III (Paclitaxel IP, Cisplatin, Bevacizumab): Six cycles of Paclitaxel 135 mg/m2 IV over 3 hours day 1, Cisplatin 75 mg/m2 IP on day 2, Paclitaxel 60 mg/m2 IP on day 8, Bevacizumab 15 mg/kg IV on day 1 beginning with cycle 2, followed by bevacizumab 15 mg/kg for cycles 7-22.
Period: Overall Study
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevcizumab IV) | Arm II (Paclitaxel,carboplatinIP, Bevacizumab IP) | Arm III (Paclitaxel IP, Cisplatin, Bevacizumab)
Started | 521 | 518 | 521
Completed | 511 | 510 | 508
Not Completed | 10 | 8 | 13
Not completed — Did not initiate study treatment | 10 | 8 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevcizumab IV) | Arm II (Paclitaxel,carboplatinIP, Bevacizumab IP) | Arm III (Paclitaxel IP, Cisplatin, Bevacizumab) | Total
Number analyzed (Participants) | 521 | 518 | 521 | 1560
Age, Customized [Count of Participants; unit: Participants]
  <40 years | 27 | 13 | 18 | 58
  40 - 49 years | 101 | 77 | 95 | 273
  50 - 59 years | 187 | 178 | 199 | 564
  60 -69 years | 152 | 181 | 151 | 484
  70 - 79 years | 51 | 64 | 53 | 168
  >79 years | 3 | 5 | 5 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 521 | 518 | 521 | 1560
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 2 | 6
  Asian | 15 | 15 | 17 | 47
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 17 | 17 | 17 | 51
  White | 473 | 478 | 476 | 1427
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 13 | 5 | 9 | 27
FIGO Stage FIGO (International Federation of Gynecology & Obstetrics) Staging [Count of Participants; unit: Participants] — FIGO staging of the Ovary was used. FIGO stage I includes all participants with disease confined to ovary. This stage has the best outcome, between 75 to 90% survival at 5 years. Stage II includes all participants with disease in ovaries and spread limited to pelvis (45 to 60% survival at 5 years). Stage III includes all participants with disease limited to abdomen. Stage IV disease includes all participants with distant metastasis outside the abdominal cavity. This stage has the worst outcome (<20% survival at 5 years)
  Participants
    Stage I-II | 56 | 56 | 51 | 163
    Stage III | 441 | 432 | 432 | 1305
    Stage IV | 24 | 30 | 38 | 92
Residual Disease Diameter [Count of Participants; unit: Participants]
  Microscopic only | 297 | 297 | 305 | 899
  0 < diameter <= 1cm | 182 | 189 | 182 | 553
  > 1cm | 42 | 32 | 34 | 108
Histology/Grade of tumor [Count of Participants; unit: Participants] — The Histology/Grade lists how many participants entered the study with each type of tumor histology and the grade for the serous tumors. Histology is the type of tissue that the tumor is comprised of. The histologic types listed below include serous, endometrioid, clear cell, mucinous and other or not specified. Grading refers to (along with staging) describes the severity. Grade 1 tumor cells look a lot like normal ovarian cells. The outcome is good for grade I tumors. Grade 2 tumors are well differentiated. Grade 3 cells are more irregular and likely to metastasize.
  Participants
    Serous/Grade1 | 20 | 12 | 27 | 59
    Serous/Grade 2 | 43 | 36 | 35 | 114
    Serous/Grade 3 | 370 | 379 | 377 | 1126
    Endometrioid | 5 | 2 | 4 | 11
    Clear Cell | 32 | 29 | 26 | 87
    Mucinous | 2 | 5 | 5 | 12
    Other/Not specified | 48 | 55 | 47 | 150

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival
Description: Estimate the median duration of progression-free survival in months. Progression is defined using Response Evaluation Criteria in Solid Tumors criteria (RECIST v1.0) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Progression-free survival is measured from date of randomization until first indication of progression based on RECIST criteria or death from any cause, or if progression-free at last contact, the date of last disease assessment up to 10 years.
Population: Intention-to-treat: All enrolled patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevcizumab IV) | Arm II (Paclitaxel,carboplatinIP, Bevacizumab IP) | Arm III (Paclitaxel IP, Cisplatin, Bevacizumab)
Number analyzed (Participants) | 521 | 518 | 521
months | 24.9 [22.3 to 27.2] | 27.3 [24.6 to 28.8] | 26.0 [23.8 to 28.0]
Statistical Analysis 1: Comparison: Arm I (Paclitaxel, Carboplatin, Bevcizumab IV) vs Arm II (Paclitaxel,carboplatinIP, Bevacizumab IP); P value.(an P value is used to determine statistical significance in a hypothesis test). from a stratified log rank test to assess equality of progression free survival hazards of arm II and arm I; Test type: Non-Inferiority or Equivalence — Study was designed to provide 80% power when arm II reduces the progression free survival event rate 20%. The critical p-value accounts for correlation between 2 primary hypotheses; p = 0.341, Log Rank — P value not adjusted for multiplicity. Significance Threshold = 0.027; Stratified by stage of disease and size of residual disease; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.81 to 1.09] — Progression free survival of arm II relative to arm I. Adjusted for stage of disease and residual size
Statistical Analysis 2: Comparison: Arm I (Paclitaxel, Carboplatin, Bevcizumab IV) vs Arm III (Paclitaxel IP, Cisplatin, Bevacizumab); P value from a log rank test comparing the progression free survival hazards of arm III to arm I; Test type: Non-Inferiority or Equivalence — Study was designed to provide 80% power when arm III reduced the true progression free survival event rate. 20% compared to arm I. Critical p value accounts for correlation between 2 primary hypotheses; p = 0.587, Log Rank — P value not adjusted for multiplicity. Significance threshold = 0.027 accounting for 2 correlated primary hypotheses; Stratified by stage of disease and size of residual disease; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.86 to 1.15] — Progression free survival hazard of arm III to arm I. Adjusted for stage of disease and residual disease size

2. Secondary Outcome: Patients With Adverse Events by Treatment Group, as Defined by NCI CTCAE (Common Terminology Criteria for Adverse Events Version 3.0) Version 3.0
Description: Eligible and treated patients. CTCAE includes grades 1-5. Grade refers to the severity of the adverse event. Grades 0 listed should be interpreted to mean there were no subjects in the arm with a toxicity to report. Grade 1 toxicities are mild; asymptomatic or mild symptoms. Grade 2 toxicities are moderate; minimal, local or noninvasive intervention indicated. Grade 3 toxicities are severe or medically significant but not immediately life-threatening. Grade 4 toxicities are life threatening. Grade 5 is death related to adverse event.
Time Frame: During treatment and up to 30 days after end of treatment
Population: Treated Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevcizumab IV) | Arm II (Paclitaxel,carboplatinIP, Bevacizumab IP) | Arm III (Paclitaxel IP, Cisplatin, Bevacizumab)
Number analyzed (Participants) | 521 | 518 | 521
Participants
  Adverse Event Grade 0 | 0 | 0 | 1
  Adverse Event Grade 1 | 1 | 0 | 0
  Adverse Event Grade 2 | 48 | 46 | 52
  Adverse Event Grade 3 | 269 | 300 | 246
  Adverse Event Grade 4 | 185 | 158 | 199
  Adverse Event Grade 5 | 8 | 6 | 10

3. Secondary Outcome: Overall Survival
Description: Estimate the median duration of overall survival in months.
Time Frame: Up to 10 years
Population: Intention-to-treat: All enrolled patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevacizumab) | Arm II (Paclitaxel, Bevacizumab, Carboplatin IP) | Arm III (Paclitaxel IP, Bevacizumab, Cisplatin IP)
Number analyzed (Participants) | 521 | 518 | 521
Months | 75.4 [67.1 to NA] — Not defined because there are insufficient number of participant with event. | 74.2 [61.9 to 78.4] | 67.6 [63.5 to 74.6]

4. Secondary Outcome: Patient Reported Quality of Life (QOL)
Description: QOL was measured with the FACT-O TOI score. Means at baseline are raw means. Scores are reported at all time points in the outcome measure table. FACT-O TOI is Trial outcome index (TOI) of the Functional assessment of cancer therapy (FACT) for ovarian cancer (FACT-O). The FACT-O TOI is composed of three subscales; Physical Well Being (PWB) ( 7 items), and Ovarian Cancer subscale (OCS) (12 items). Each item in the FACT-O TOI are scored using a 5 point scale (0=not at all; 1=a little bit; 2=somewhat;3=quite a bit;4=very much). A subscale score is computed as long as more thatn 50% of subscale items have been answered. A total score of the FACT-O items provide valid responses and all three subscales have valid scores. A score of the FACT-) TOI is ranged 0-104 with a larger score indicating a more preferred state of health-related quality of life (HRQOL).
Time Frame: Time points: Baseline, prior to cycle 4, prior to cycle 7, prior to cycle 13, prior to cycle 21, up to 84 weeks post starting treatment
Population: Patients evaluable for PRO (Patient Reported Outcomes)/QOL (completed baseline and at least one follow-up assessment)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevacizumab) | Arm II (Paclitaxel, Bevacizumab, Carboplatin IP) | Arm III (Paclitaxel IP, Bevacizumab, Cisplatin IP)
Number analyzed (Participants) | 492 | 481 | 464
Units on a scale
  Baseline | 68.5 (0.7) | 67.4 (0.7) | 67.7 (0.7)
  Prior to cycle 4 | 67.8 (0.6) | 65.6 (0.6) | 61.9 (0.6)
  Prior to cycle 7 | 69.1 (0.6) | 68.2 (0.6) | 65.7 (0.7)
  Prior to cycle 13 | 77.3 (0.6) | 77.1 (0.6) | 78.4 (0.6)
  Prior to cycle 21 | 77.7 (0.6) | 76.9 (0.7) | 78.2 (0.6)
  84 weeks | 78.3 (0.7) | 77.7 (0.7) | 79.4 (0.7)

5. Secondary Outcome: Patient Reported Neurotoxicity (Ntx)
Description: The FACT/GOG-NTX subscale (short version) contains 4 items measuring sensory neuropathy. Each item is scored using a 5 point Likert scale (0=not at all; 1=a little bit;2=somewhat;3=quite a bit; 4=very much). For each item, reversal was performed prior to score calculation so that a large score suggests less symptoms. According to the FACIT measurement system, the subscale score was calculated as the summation of the individual item scores if more than 50% of a subscale items were answered. When unanswered items existed, a subscale score was prorated by multiplying the mean of the answered item scores by the number of items in the subscale. The Ntx subscale score ranges from 0-16 with a large subscale score suggesting less symptom or better QOL.
Time Frame: Time points: Baseline, prior to cycle 4, prior to cycle 7, prior to cycle 13, prior to cycle 21, 84 weeks post starting treatment
Population: Patients evaluable for PRO(Patient Reported Outcome)/QOL (completed baseline and at least one follow-up assessment).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevacizumab) | Arm II (Paclitaxel, Bevacizumab, Carboplatin IP) | Arm III (Paclitaxel IP, Bevacizumab, Cisplatin IP)
Number analyzed (Participants) | 492 | 481 | 464
Units on a scale
  Baseline | 15.4 (0.1) | 15.4 (0.1) | 15.4 (0.1)
  Prior to cycle 4 | 12.9 (0.2) | 13.0 (0.2) | 13.6 (0.2)
  Prior to cycle 7 | 10.4 (0.2) | 10.3 (0.2) | 10.9 (0.2)
  Prior to cycle 13 | 11.1 (0.2) | 10.5 (0.2) | 9.2 (0.2)
  Prior to cycle 21 | 11.4 (0.2) | 11.1 (0.2) | 11.0 (0.2)
  84 weeks | 11.9 (0.2) | 11.4 (0.2) | 11.5 (0.2)

6. Secondary Outcome: Patient Reported Fatigue
Description: Patient reported fatigue as measured with the Functional Assessment of Chronic Illness Therapy- Fatigue scale (FACIT-Fatigue). The FACIT-Fatigue contains 13 items. Each item was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). For the negative items, reversal was performed prior to score calculation. According to the FACIT measurement system, the Fatigue score was the summation of the individual item scores if more than 50% of subscale items were answered. When unanswered items existed, a subscale score was prorated by multiplying the mean of the answered item scores by the number of items in the scale. The FACIT-Fatigue score ranges 0-52 with a large score suggesting less fatigue.
Time Frame: as for outcome 5
Population: Patients evaluable for PRO (Patient Reported Outcomes)/QOL. Evaluable patients have completed baseline and at least one follow-up assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevacizumab) | Arm II (Paclitaxel, Bevacizumab, Carboplatin IP) | Arm III (Paclitaxel IP, Bevacizumab, Cisplatin IP)
Number analyzed (Participants) | 492 | 481 | 464
units on a scale
  Baseline | 35.3 (0.3) | 35.1 (0.3) | 35.3 (0.3)
  Prior to cycle 4 | 32.5 (0.3) | 32.0 (0.3) | 31.3 (0.3)
  Prior to cycle 7 | 32.7 (0.3) | 32.7 (0.3) | 32.4 (0.3)
  Prior to cycle 13 | 35.7 (0.3) | 35.5 (0.3) | 35.9 (0.3)
  Prior to cycle 21 | 35.5 (0.3) | 35.1 (0.3) | 36.3 (0.3)
  84 weeks | 35.7 (0.3) | 36.0 (0.3) | 36.5 (0.3)

7. Secondary Outcome: Patient Reported Nausea
Description: Nausea was measured with the a single item ,' I have nausea' from the FACT-O TOI, and was scored using a 5 point scale (0=not at all; 1=a little bit; 2=somewhat;3=quite a bit;4=very much)
Time Frame: as for outcome 5
Population: Patients evaluable for PRO (Patient Reported Outcomes)/QOL are patients who completed baseline and at least one follow-up assessment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevacizumab) | Arm II (Paclitaxel, Bevacizumab, Carboplatin IP) | Arm III (Paclitaxel IP, Bevacizumab, Cisplatin IP)
Number analyzed (Participants) | 492 | 481 | 464
units on a scale
  Baseline | 0.4 (0.04) | 0.4 (0.04) | 0.4 (0.04)
  Prior to cycle 4 | 0.6 (0.04) | 0.7 (0.04) | 1.1 (0.05)
  Prior to cycle 7 | 0.5 (0.04) | 0.5 (0.04) | 0.7 (0.05)
  Prior to cycle 13 | 0.2 (0.03) | 0.3 (0.03) | 0.2 (0.03)
  Prior to cycle 21 | 0.3 (0.04) | 0.4 (0.04) | 0.3 (0.03)
  84 Weeks | 0.3 (0.04) | 0.4 (0.04) | 0.3 (0.03)

ADVERSE EVENTS:
Time Frame: AEs were recorded from the initiation of any study treatment up until 30 days following the last cycle of study treatment.
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevcizumab IV) | Arm II (Paclitaxel,carboplatinIP, Bevacizumab IP) | Arm III (Paclitaxel IP, Cisplatin, Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 156/511 | 179/510 | 215/508
Other Adverse Events (participants affected / at risk) | 511/511 | 510/510 | 507/508
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel, Carboplatin, Bevcizumab IV) (N=511) | Arm II (Paclitaxel,carboplatinIP, Bevacizumab IP) (N=510) | Arm III (Paclitaxel IP, Cisplatin, Bevacizumab) (N=508)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 2 | 2 | 2
Neutrophils (Blood and lymphatic system disorders) | 10 | 6 | 4
Platelets (Blood and lymphatic system disorders) | 2 | 1 | 0
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytes (Blood and lymphatic system disorders) | 1 | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 1 | 2 | 0
Sinus/Node (S/N) Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 2 | 2 | 3
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 2
Cardiac Ischemia/Infarction (Cardiac disorders) | 2 | 4 | 1
Right Ventricular Dysfunction (Cardiac disorders) | 0 | 0 | 1
Hypertension (Cardiac disorders) | 4 | 5 | 12
Restrictive Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Left Venticular Diastolic Dysfunction (Cardiac disorders) | 0 | 1 | 0
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 0 | 0 | 1
Cardiac General - Other (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
International Normalized ratio (Inr) (Vascular disorders) | 1 | 0 | 0
Fever (General disorders) | 1 | 2 | 4
Weight Loss (General disorders) | 1 | 0 | 0
Rigors/Chills (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 2 | 1
Death No Ctcae Term - Disease Progression Not otherwise specified (NOS) (General disorders) | 2 | 0 | 1
Death No Ctcae Term - Death Nos (General disorders) | 0 | 1 | 0
Death No Ctcae Term - Multi-Organ Failure (General disorders) | 1 | 0 | 1
Death No Ctcae Term - Sudden Death (General disorders) | 0 | 0 | 3
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 2 | 7 | 5
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Fistula, Gi - Colon/Cecum/Appendix (Gastrointestinal disorders) | 1 | 1 | 2
Enteritis (Gastrointestinal disorders) | 1 | 1 | 0
Perforation, Gastrointestinal (GI) - Duodenum (Gastrointestinal disorders) | 1 | 0 | 0
Perforation, Gi - Appendix (Gastrointestinal disorders) | 1 | 0 | 0
Obstruction, Gi - Ileum (Gastrointestinal disorders) | 0 | 2 | 0
Necrosis, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1 | 0 | 0
Perforation, Gi - Colon (Gastrointestinal disorders) | 5 | 2 | 4
Fistula, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1 | 3 | 2
Fistula, Gi - Rectum (Gastrointestinal disorders) | 2 | 0 | 0
Obstruction, Gi - Colon (Gastrointestinal disorders) | 1 | 1 | 2
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Leak, Gi - Large Bowel (Gastrointestinal disorders) | 1 | 1 | 0
Leak, Gi - Leak Nos (Gastrointestinal disorders) | 1 | 0 | 0
Fistula, Gi - Anus (Gastrointestinal disorders) | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 2 | 3 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Distention (Gastrointestinal disorders) | 0 | 0 | 1
Fistula, Gi - Abdomen Nos (Gastrointestinal disorders) | 0 | 1 | 0
Obstruction, Gi - Gallbladder (Gastrointestinal disorders) | 0 | 1 | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 0 | 0 | 2
Obstruction, Gi - Duodenal (Gastrointestinal disorders) | 0 | 1 | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 17 | 20 | 12
Colitis (Gastrointestinal disorders) | 0 | 1 | 1
Obstruction, Gi - Jejunum (Gastrointestinal disorders) | 3 | 0 | 0
Perforation, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1 | 2 | 4
Vomiting (Gastrointestinal disorders) | 2 | 2 | 13
Dehydration (Gastrointestinal disorders) | 1 | 7 | 9
Constipation (Gastrointestinal disorders) | 2 | 1 | 6
Nausea (Gastrointestinal disorders) | 1 | 3 | 5
Gastrointestinal - Other (Gastrointestinal disorders) | 0 | 2 | 3
Perforation, Gi - Ileum (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 5
Hemorrhage, Genitourinary (Gu) - Urinary Nos (Vascular disorders) | 1 | 0 | 0
Hemorrhage, Gu - Vagina (Vascular disorders) | 0 | 0 | 1
Hemorrhage, Gi - Rectum (Vascular disorders) | 0 | 2 | 1
Hemorrhage, Gi - Peritoneal Cavity (Vascular disorders) | 1 | 0 | 0
Hemorrhage, Gi - Upper Gi Nos (Vascular disorders) | 2 | 0 | 1
Hemorrhage With Surgery (Vascular disorders) | 1 | 0 | 0
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 0 | 3 | 3
Hematoma (Vascular disorders) | 1 | 2 | 1
Hemorrhage, Gi - Lower Gi Nos (Vascular disorders) | 0 | 1 | 0
Hemorrhage, Gi - Stomach (Vascular disorders) | 0 | 0 | 1
Hemorrhage, Gi - Colon (Vascular disorders) | 1 | 0 | 0
Hemorrhage, Cns (Vascular disorders) | 0 | 0 | 3
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Pancreatitis (Hepatobiliary disorders) | 0 | 0 | 3
Infection (Inf) with Grade 3 Or 4 Absolute Neutrophil Count (Anc): Wound (Infections and infestations) | 1 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 2 | 1 | 1
Inf W/Gr 3 Or 4 Anc: Colon (Infections and infestations) | 0 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Anal/Perianal (Infections and infestations) | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Skin (Cellulitis) (Infections and infestations) | 0 | 1 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Mediastinum Nos (Infections and infestations) | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 3 | 2 | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Gallbladder (Infections and infestations) | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 0 | 2 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 2 | 4 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Appendix (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 3 | 1 | 5
Inf W/Nml Or Gr 1 Or 2 Anc: Catheter-Related (Infections and infestations) | 2 | 3 | 7
Febrile Neutropenia (Infections and infestations) | 6 | 4 | 7
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Dental-Tooth (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Colon (Infections and infestations) | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 1 | 4 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 0 | 3 | 3
Inf Unknown Anc: Blood (Infections and infestations) | 1 | 1 | 2
Infection - Other (Infections and infestations) | 2 | 2 | 2
Opportunisitic Inf Assoc. W/Gr 2 Lymphopenia (Infections and infestations) | 0 | 1 | 0
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 0 | 1 | 4
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 1 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Abdomen Nos (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Up. Aerodigestive (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Pelvis Nos (Infections and infestations) | 0 | 5 | 0
Inf W/Nml Or Gr 1 Or 2 Anc:peritoneal Cavity (Infections and infestations) | 0 | 1 | 1
Inf Unknown Anc: Catheter-Related (Infections and infestations) | 1 | 0 | 1
Inf Unknown Anc: Rectum (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Foreign Body (Infections and infestations) | 1 | 0 | 0
Inf Unknown Anc: Abdomen Nos (Infections and infestations) | 0 | 0 | 1
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 0 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Upper Airway Nos (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Anal/Perianal (Infections and infestations) | 1 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Lung (Pneumonia) (Infections and infestations) | 1 | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 2 | 1 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 0 | 1 | 1
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 0 | 2 | 2
Inf W/Gr 3 Or 4 Anc: Catheter-Related (Infections and infestations) | 1 | 0 | 1
Lymphocele (Blood and lymphatic system disorders) | 0 | 1 | 1
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 0 | 1 | 0
Proteinuria (Metabolism and nutrition disorders) | 1 | 2 | 1
Creatinine (Metabolism and nutrition disorders) | 1 | 1 | 4
Alanine Aminotransferase (Alt) (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 2
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Seroma (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Device/Prosthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle Weakness - Extremity-Upper (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 5 | 1 | 7
Neurology - Other (Nervous system disorders) | 0 | 1 | 2
Encephalopathy (Nervous system disorders) | 1 | 0 | 1
Mood Alteration - Anxiety (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Speech Impairment (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 4
Personality (Nervous system disorders) | 1 | 0 | 1
Cognitive Disturbance (Nervous system disorders) | 0 | 0 | 1
Central Nervous System (Cns) Ischemia (Nervous system disorders) | 2 | 2 | 4
Confusion (Nervous system disorders) | 1 | 1 | 0
Memory Impairment (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Neuropathy-Sensory (Nervous system disorders) | 3 | 2 | 0
Blurred Vision (Eye disorders) | 1 | 0 | 0
Pain - Other (General disorders) | 0 | 1 | 0
Pain: Chest /Thorax Nos (General disorders) | 0 | 0 | 1
Pain: Head/Headache (General disorders) | 1 | 1 | 2
Pain: Neck (General disorders) | 0 | 0 | 2
Pain: Joint (General disorders) | 0 | 0 | 1
Pain: Bladder (General disorders) | 0 | 1 | 0
Pain: Oral Cavity (General disorders) | 0 | 1 | 0
Pain: Esophagus (General disorders) | 1 | 1 | 0
Pain: Abdominal Pain Nos (General disorders) | 6 | 13 | 12
Pain: Cardiac/ Heart (General disorders) | 0 | 0 | 1
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 2
Renal/Genitourinary - Other (Renal and urinary disorders) | 3 | 0 | 0
Perforation, Gu - Vagina (Renal and urinary disorders) | 1 | 0 | 0
Leak, Gu - Vagina (Renal and urinary disorders) | 0 | 1 | 0
Urinary Color Change (Renal and urinary disorders) | 0 | 1 | 0
Obstruction, Gu - Ureter (Renal and urinary disorders) | 0 | 0 | 1
Fistula, Gu - Vagina (Renal and urinary disorders) | 0 | 1 | 1
Fistula, Gu - Bladder (Renal and urinary disorders) | 0 | 2 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 1
2nd Malignancy: Poss. Related To Cancer Rx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Syndromes - Other (General disorders) | 0 | 1 | 3
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 0 | 1 | 0
Thrombosis/Thrombus/Embolism (Vascular disorders) | 25 | 25 | 25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel, Carboplatin, Bevcizumab IV) (N=511) | Arm II (Paclitaxel,carboplatinIP, Bevacizumab IP) (N=510) | Arm III (Paclitaxel IP, Cisplatin, Bevacizumab) (N=508)
Allergy/Immunology - Other (Immune system disorders) | 3 | 1 | 1
Allergic Reaction/Hypersensitivity (Immune system disorders) | 36 | 51 | 54
Vasculitis (Immune system disorders) | 0 | 1 | 1
Rhinitis (Immune system disorders) | 141 | 119 | 103
Autoimmune Reaction (Immune system disorders) | 1 | 2 | 0
Otitis Middle Ear (Ear and labyrinth disorders) | 6 | 1 | 1
Auditory/Ear - Other (Ear and labyrinth disorders) | 1 | 2 | 1
Otitis External Ear (Ear and labyrinth disorders) | 0 | 2 | 2
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 12 | 9 | 21
Tinnitus (Ear and labyrinth disorders) | 60 | 33 | 59
Hearing (Monitoring Program) (Ear and labyrinth disorders) | 5 | 2 | 6
Neutrophils (Blood and lymphatic system disorders) | 484 | 473 | 462
Platelets (Blood and lymphatic system disorders) | 371 | 370 | 253
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 3 | 1 | 4
Leukocytes (Blood and lymphatic system disorders) | 486 | 480 | 459
Lymphopenia (Blood and lymphatic system disorders) | 48 | 55 | 44
Hemolysis (Blood and lymphatic system disorders) | 1 | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 499 | 490 | 483
Prolonged Q wave and tc wave Interval (Cardiac disorders) | 0 | 1 | 1
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 2 | 1 | 2
Conduction Abnml: Conduction Abnormality Nos (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 41 | 25 | 31
Cardiac Arrhythmia - Other (Cardiac disorders) | 3 | 0 | 0
Conduction Abnml: Av Block 1st Degree (Cardiac disorders) | 0 | 1 | 0
Ventricular Arrhythmia - Tachycardia (Cardiac disorders) | 5 | 5 | 3
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 26 | 20 | 15
Vasovagal Episode (Cardiac disorders) | 0 | 2 | 4
Supraventricular Tachycardia (Cardiac disorders) | 3 | 4 | 3
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 1 | 1 | 7
Ventricular Arrhythmia - Pvcs (Cardiac disorders) | 1 | 2 | 0
Ventricular Arrhythmia - Trigeminny (Cardiac disorders) | 1 | 0 | 0
Ventricular Arrhythmia - Bigeminy (Cardiac disorders) | 2 | 0 | 0
S/N Arrhythmia: Atrial Tachycardia (Cardiac disorders) | 2 | 0 | 0
Cardiac Ischemia/Infarction (Cardiac disorders) | 1 | 0 | 1
Right Ventricular Dysfunction (Cardiac disorders) | 1 | 0 | 1
Pulmonary Hypertension (Cardiac disorders) | 1 | 1 | 0
Hypertension (Cardiac disorders) | 205 | 189 | 242
Valvular Heart Disease (Cardiac disorders) | 2 | 0 | 0
Left Venticular Diastolic Dysfunction (Cardiac disorders) | 1 | 0 | 1
Lt Ventricular Systolic Dysfunction (Cardiac disorders) | 0 | 2 | 1
Cardiac General - Other (Cardiac disorders) | 0 | 0 | 1
Cardiac Troponin I (Ctni) (Cardiac disorders) | 1 | 2 | 1
Cardiac Troponin T (Ctnt) (Cardiac disorders) | 0 | 1 | 1
Pericardial Effusion (Cardiac disorders) | 1 | 0 | 1
Hypotension (Cardiac disorders) | 15 | 19 | 29
Inr (Vascular disorders) | 12 | 10 | 16
Partial Throboplastin Time (Ptt) (Vascular disorders) | 10 | 10 | 12
Constitutional Symptoms - Other (General disorders) | 6 | 2 | 2
Sweating (General disorders) | 25 | 19 | 23
Weight Gain (General disorders) | 121 | 105 | 82
Patient Odor (General disorders) | 0 | 0 | 1
Fever (General disorders) | 55 | 68 | 62
Weight Loss (General disorders) | 64 | 80 | 97
Hypothermia (General disorders) | 0 | 0 | 1
Rigors/Chills (General disorders) | 24 | 26 | 37
Fatigue (General disorders) | 465 | 457 | 451
Insomnia (General disorders) | 160 | 151 | 150
Death No Ctcae Term - Death Nos (General disorders) | 0 | 1 | 0
Nail Changes (Skin and subcutaneous tissue disorders) | 137 | 113 | 48
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 7 | 11 | 19
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 402 | 378 | 377
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 3 | 2 | 1
Dermatitis - Chemoradiation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypopigmentation (Skin and subcutaneous tissue disorders) | 4 | 4 | 3
Induration (Skin and subcutaneous tissue disorders) | 2 | 9 | 3
Cheilitis (Skin and subcutaneous tissue disorders) | 3 | 1 | 2
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 34 | 43 | 46
Bruising (Skin and subcutaneous tissue disorders) | 43 | 49 | 31
Acne (Skin and subcutaneous tissue disorders) | 5 | 13 | 16
Rash (Skin and subcutaneous tissue disorders) | 186 | 192 | 121
Dry Skin (Skin and subcutaneous tissue disorders) | 61 | 51 | 29
Decubitus (Skin and subcutaneous tissue disorders) | 0 | 2 | 4
Atrophy, Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 43 | 39 | 36
Burn (Skin and subcutaneous tissue disorders) | 4 | 6 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 4 | 2
Flushing (Skin and subcutaneous tissue disorders) | 30 | 26 | 25
Hand-Foot (Skin and subcutaneous tissue disorders) | 13 | 11 | 6
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 17 | 24 | 9
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 15 | 20 | 8
Ulceration (Skin and subcutaneous tissue disorders) | 8 | 13 | 4
Hot Flashes (Endocrine disorders) | 103 | 84 | 89
Diabetes (Endocrine disorders) | 2 | 1 | 0
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 1
Adrenal Insufficiency (Endocrine disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 1 | 1
Endocrine - Other (Endocrine disorders) | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 7 | 10 | 4
Cushingoid (Endocrine disorders) | 2 | 3 | 0
Fistula, Gi - Colon/Cecum/Appendix (Gastrointestinal disorders) | 0 | 4 | 1
Enteritis (Gastrointestinal disorders) | 2 | 4 | 0
Perforation, Gi - Duodenum (Gastrointestinal disorders) | 0 | 0 | 1
Ulcer,gi - Colon (Gastrointestinal disorders) | 1 | 0 | 0
Obstruction, Gi - Ileum (Gastrointestinal disorders) | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 3 | 0 | 0
Ulcer,gi - Anus (Gastrointestinal disorders) | 1 | 1 | 0
Salivary Gland Changes (Gastrointestinal disorders) | 1 | 0 | 6
Flatulence (Gastrointestinal disorders) | 24 | 22 | 26
Perforation, Gi - Colon (Gastrointestinal disorders) | 0 | 0 | 2
Ulcer,gi - Duodenum (Gastrointestinal disorders) | 0 | 1 | 1
Fistula, Gi - Ileum (Gastrointestinal disorders) | 1 | 1 | 0
Dental: Periodontal (Gastrointestinal disorders) | 6 | 6 | 2
Fistula, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1 | 3 | 0
Fistula, Gi - Rectum (Gastrointestinal disorders) | 3 | 0 | 0
Obstruction, Gi - Colon (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 9 | 7 | 10
Ulcer,gi - Stoma (Gastrointestinal disorders) | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 7 | 5 | 9
Hemorrhoids (Gastrointestinal disorders) | 45 | 38 | 24
Heartburn (Gastrointestinal disorders) | 97 | 80 | 107
Ulcer,gi - Stomach (Gastrointestinal disorders) | 2 | 3 | 1
Dental: Teeth (Gastrointestinal disorders) | 11 | 10 | 12
Mucositis (Functional/Sympt) - Pharynx (Gastrointestinal disorders) | 4 | 1 | 0
Fistula, Gi - Jejunum (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 10 | 5
Fistula, Gi - Anus (Gastrointestinal disorders) | 0 | 2 | 3
Leak, Gi - Rectum (Gastrointestinal disorders) | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 2 | 5 | 3
Dental: Teeth Development (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 23 | 23 | 21
Distention (Gastrointestinal disorders) | 47 | 63 | 93
Taste Alteration (Gastrointestinal disorders) | 117 | 100 | 97
Incontinence, Anal (Gastrointestinal disorders) | 1 | 5 | 5
Fistula, Gi - Abdomen Nos (Gastrointestinal disorders) | 0 | 4 | 1
Dry Mouth (Gastrointestinal disorders) | 22 | 17 | 15
Mucositis (Functional/Sympt) - Stomach (Gastrointestinal disorders) | 1 | 1 | 1
Obstruction, Gi - Gallbladder (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis (Functional/Sympt) - Rectum (Gastrointestinal disorders) | 0 | 1 | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 89 | 80 | 48
Stricture, Gi - Colon (Gastrointestinal disorders) | 1 | 0 | 0
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 3 | 5 | 6
Fistula, Gi - Oral Cavity (Gastrointestinal disorders) | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 4 | 4 | 5
Mucositis (Clinical Exam) - Stomach (Gastrointestinal disorders) | 1 | 0 | 2
Mucositis (Functional/Sympt) - Anus (Gastrointestinal disorders) | 0 | 1 | 0
Perforation, Gi - Small Bowel Nos (Gastrointestinal disorders) | 2 | 1 | 0
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 117 | 107 | 76
Mucositis (Clinical Exam) - Larynx (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis (Clinical Exam) - Esophagus (Gastrointestinal disorders) | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 158 | 160 | 215
Anorexia (Gastrointestinal disorders) | 161 | 159 | 211
Dehydration (Gastrointestinal disorders) | 26 | 52 | 93
Constipation (Gastrointestinal disorders) | 321 | 323 | 335
Stricture, Gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 317 | 331 | 393
Malabsorption (Gastrointestinal disorders) | 0 | 2 | 0
Gastrointestinal - Other (Gastrointestinal disorders) | 11 | 9 | 10
Perforation, Gi - Ileum (Gastrointestinal disorders) | 0 | 0 | 1
Leak, Gi - Stomach (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 224 | 263 | 264
Prolapse Of Stoma, Gi (Gastrointestinal disorders) | 2 | 2 | 0
Mucositis (Clinical Exam) - Pharynx (Gastrointestinal disorders) | 3 | 0 | 2
Perforation, Gi - Jejunum (Gastrointestinal disorders) | 0 | 0 | 1
Hemorrhage, Gu - Stoma (Vascular disorders) | 0 | 1 | 1
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 6 | 5 | 4
Hemorrhage, Gu - Vagina (Vascular disorders) | 16 | 21 | 9
Hemorrhage/Pulmonary - Bronchopulmonary Nos (Vascular disorders) | 3 | 1 | 1
Hemorrhage/Pulmonary - Lung (Vascular disorders) | 0 | 1 | 2
Hemorrhage/Pulmonary - Pharynx (Vascular disorders) | 1 | 1 | 0
Hemorrhage, Gi - Rectum (Vascular disorders) | 36 | 23 | 15
Hemorrhage/Pulmonary - Respiratory Tract Nos (Vascular disorders) | 2 | 3 | 1
Hemorrhage, Gi - Stoma (Vascular disorders) | 2 | 0 | 0
Hemorrhage, Gi - Varices (Rectal) (Vascular disorders) | 3 | 1 | 3
Hemorrhage, Gi - Peritoneal Cavity (Vascular disorders) | 0 | 0 | 1
Hemorrhage, Gi - Upper Gi Nos (Vascular disorders) | 1 | 1 | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 261 | 231 | 184
Hematoma (Vascular disorders) | 2 | 8 | 11
Hemorrhage, Gi - Anus (Vascular disorders) | 8 | 12 | 5
Hemorrhage, Gi - Esophagus (Vascular disorders) | 0 | 1 | 0
Hemorrhage, Gu - Ureter (Vascular disorders) | 0 | 1 | 0
Hemorrhage, Gi - Duodenum (Vascular disorders) | 1 | 0 | 0
Hemorrhage, Gi - Lower Gi Nos (Vascular disorders) | 4 | 2 | 5
Hemorrhage, Gi - Oral Cavity (Vascular disorders) | 38 | 32 | 26
Hemorrhage, Gu - Kidney (Vascular disorders) | 1 | 0 | 0
Hemorrhage, Gu - Bladder (Vascular disorders) | 3 | 1 | 4
Hemorrhage, Gi - Stomach (Vascular disorders) | 1 | 0 | 0
Hemorrhage, Gi - Colon (Vascular disorders) | 2 | 0 | 1
Hemorrhage, Cns (Vascular disorders) | 0 | 3 | 4
Petechiae (Vascular disorders) | 9 | 2 | 3
Hemorrhage/Bleeding - Other (Vascular disorders) | 2 | 2 | 3
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 3
Liver Dysfunction (Hepatobiliary disorders) | 3 | 0 | 0
Pancreatitis (Hepatobiliary disorders) | 1 | 2 | 1
Inf W/Gr 3 Or 4 Anc: Wound (Infections and infestations) | 2 | 2 | 3
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 2 | 3 | 2
Inf W/Gr 3 Or 4 Anc: Foreign Body (Infections and infestations) | 0 | 2 | 0
Inf W/Gr 3 Or 4 Anc: Dental-Tooth (Infections and infestations) | 1 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Colon (Infections and infestations) | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Anal/Perianal (Infections and infestations) | 1 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Ungual (Nails) (Infections and infestations) | 0 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Skin (Cellulitis) (Infections and infestations) | 4 | 3 | 2
Inf W/Gr 3 Or 4 Anc: Middle Ear (Infections and infestations) | 0 | 1 | 0
Inf W/Gr 3 Or 4 Anc: External Ear (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Vulva (Infections and infestations) | 0 | 2 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 24 | 32 | 28
Inf W/Nml Or Gr 1 Or 2 Anc: Paranasal (Infections and infestations) | 2 | 2 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Nose (Infections and infestations) | 2 | 0 | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Neck Nos (Infections and infestations) | 1 | 0 | 0
Infection (Inf) With Normal Or Grade 1 Or 2 Absolute Neutrophil Count (Anc): Mediastinum Nos (Infections and infestations) | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 7 | 8 | 4
Inf W/Nml Or Gr 1 Or 2 Anc: Larynx (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Eye Nos (Infections and infestations) | 1 | 1 | 4
Inf W/Gr 3 Or 4 Anc: Peritoneal Cavity (Infections and infestations) | 2 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Small Bowel Nos (Infections and infestations) | 0 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Esophagus (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Soft Tissue Nos (Infections and infestations) | 0 | 2 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Joint (Infections and infestations) | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Biliary Tree (Infections and infestations) | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urethra (Infections and infestations) | 1 | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 2 | 3 | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 9 | 16 | 17
Inf W/Nml Or Gr 1 Or 2 Anc: Small Bowel Nos (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Oral Cavity-Gums (Infections and infestations) | 4 | 6 | 4
Inf W/Nml Or Gr 1 Or 2 Anc: Otitis Media Nos (Infections and infestations) | 2 | 1 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 13 | 22 | 17
Inf W/Nml Or Gr 1 Or 2 Anc: Catheter-Related (Infections and infestations) | 9 | 10 | 13
Febrile Neutropenia (Infections and infestations) | 7 | 10 | 11
Inf W/Nml Or Gr 1 Or 2 Anc: Lip/Perioral (Infections and infestations) | 1 | 1 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Rectum (Infections and infestations) | 0 | 1 | 0
Infection (Inf) Unknown Absolute Neutrophil Count (Anc): Lung (Pneumonia) (Infections and infestations) | 0 | 1 | 3
Inf Unknown Anc: Nose (Infections and infestations) | 1 | 0 | 0
Inf Unknown Anc: Sinus (Infections and infestations) | 16 | 7 | 11
Inf W/Nml Or Gr 1 Or 2 Anc: Dental-Tooth (Infections and infestations) | 8 | 3 | 5
Inf W/Nml Or Gr 1 Or 2 Anc: Colon (Infections and infestations) | 1 | 1 | 1
Viral Hepatitis (Infections and infestations) | 1 | 2 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 40 | 42 | 46
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 5 | 6 | 6
Inf W/Nml Or Gr 1 Or 2 Anc: Ungual (Nails) (Infections and infestations) | 12 | 13 | 2
Inf Unknown Anc: Blood (Infections and infestations) | 0 | 1 | 0
Inf Unknown Anc: Stomach (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Stomach (Infections and infestations) | 1 | 3 | 1
Infection - Other (Infections and infestations) | 16 | 12 | 12
Inf W/Gr 3 Or 4 Anc: Bladder (Urinary) (Infections and infestations) | 5 | 4 | 1
Opportunisitic Inf Assoc. W/Gr 2 Lymphopenia (Infections and infestations) | 2 | 2 | 1
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 4 | 9 | 4
Inf W/Nml Or Gr 1 Or 2 Anc: Nerve-Peripheral (Infections and infestations) | 0 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Oral Cavity-Gums (Infections and infestations) | 0 | 3 | 1
Inf Unknown Anc: Vulva (Infections and infestations) | 1 | 1 | 0
Inf Unknown Anc: Vagina (Infections and infestations) | 1 | 3 | 6
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 6 | 8 | 4
Inf W/Gr 3 Or 4 Anc: Abdomen Nos (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Mucosa (Infections and infestations) | 0 | 1 | 0
Inf Unknown Anc: Pelvis Nos (Infections and infestations) | 1 | 2 | 0
Inf Unknown Anc: Upper Airway Nos (Infections and infestations) | 12 | 12 | 9
Inf Unknown Anc: Upper Aerodigestive (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Pharynx (Infections and infestations) | 5 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Vagina (Infections and infestations) | 8 | 7 | 9
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 25 | 27 | 18
Inf W/Nml Or Gr 1 Or 2 Anc: Pelvis Nos (Infections and infestations) | 1 | 4 | 2
Inf Unknown Anc: Pharynx (Infections and infestations) | 0 | 1 | 2
Inf Unknown Anc: Mucosa (Infections and infestations) | 0 | 1 | 1
Inf Unknown Anc: Bronchus (Infections and infestations) | 4 | 2 | 3
Inf Unknown Anc: Eye Nos (Infections and infestations) | 2 | 0 | 1
Inf Unknown Anc: Nerve-Cranial (Infections and infestations) | 0 | 1 | 0
Inf Unknown Anc: Soft Tissue Nos (Infections and infestations) | 0 | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc:peritoneal Cavity (Infections and infestations) | 1 | 1 | 4
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 16 | 26 | 11
Inf Unknown Anc: Urethra (Infections and infestations) | 0 | 1 | 0
Inf Unknown Anc: Bladder (Urinary) (Infections and infestations) | 6 | 14 | 5
Inf Unknown Anc: Wound (Infections and infestations) | 0 | 2 | 1
Inf Unknown Anc: Foreign Body (Infections and infestations) | 1 | 0 | 0
Inf Unknown Anc: Catheter-Related (Infections and infestations) | 1 | 4 | 5
Inf Unknown Anc: Rectum (Infections and infestations) | 0 | 1 | 0
Inf Unknown Anc: Peritoneal Cavity (Infections and infestations) | 0 | 1 | 1
Inf Unknown Anc: Oral Cavity-Gums (Infections and infestations) | 1 | 2 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Foreign Body (Infections and infestations) | 1 | 0 | 3
Inf Unknown Anc: Dental-Tooth (Infections and infestations) | 5 | 3 | 7
Inf Unknown Anc: Colon (Infections and infestations) | 0 | 1 | 1
Inf Unknown Anc: Appendix (Infections and infestations) | 0 | 1 | 0
Inf Unknown Anc: Anal/Perianal (Infections and infestations) | 2 | 1 | 0
Inf Unknown Anc: Abdomen Nos (Infections and infestations) | 0 | 1 | 4
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 9 | 9 | 4
Inf Unknown Anc: Lip/Perioral (Infections and infestations) | 0 | 0 | 2
Inf Unknown Anc: Middle Ear (Infections and infestations) | 2 | 1 | 0
Inf Unknown Anc: External Ear (Infections and infestations) | 1 | 0 | 3
Inf W/Gr 3 Or 4 Anc: Vagina (Infections and infestations) | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Upper Airway Nos (Infections and infestations) | 0 | 2 | 0
Inf W/Gr 3 Or 4 Anc: Upper Aerodigestive (Infections and infestations) | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Anal/Perianal (Infections and infestations) | 5 | 5 | 3
Inf W/Gr 3 Or 4 Anc: Sinus (Infections and infestations) | 4 | 2 | 2
Inf W/Gr 3 Or 4 Anc: Nose (Infections and infestations) | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Mucosa (Infections and infestations) | 0 | 2 | 1
Inf W/Gr 3 Or 4 Anc: Lung (Pneumonia) (Infections and infestations) | 0 | 1 | 1
Inf W/Gr 3 Or 4 Anc: Eye Nos (Infections and infestations) | 1 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Conjunctiva (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 0 | 1 | 1
Inf Unknown Anc: Ungual (Nails) (Infections and infestations) | 3 | 5 | 1
Inf W/Gr 3 Or 4 Anc: Soft Tissue Nos (Infections and infestations) | 1 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Lymphatic (Infections and infestations) | 2 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 11 | 7 | 4
Inf Unknown Anc: Esophagus (Infections and infestations) | 0 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 4 | 11 | 7
Inf W/Nml Or Gr 1 Or 2 Anc: External Ear (Infections and infestations) | 2 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Urethra (Infections and infestations) | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Catheter-Related (Infections and infestations) | 0 | 3 | 0
Inf W/Gr 3 Or 4 Anc: Kidney (Infections and infestations) | 1 | 0 | 0
Lymphedema-Related Fibrosis (Blood and lymphatic system disorders) | 1 | 0 | 3
Lymphatics - Other (Blood and lymphatic system disorders) | 1 | 2 | 1
Lymphocele (Blood and lymphatic system disorders) | 6 | 4 | 3
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 8 | 4 | 9
Edema: Limb (Blood and lymphatic system disorders) | 101 | 106 | 94
Edema: Head And Neck (Blood and lymphatic system disorders) | 12 | 5 | 10
Dermal Change (Blood and lymphatic system disorders) | 0 | 1 | 1
Ast (Metabolism and nutrition disorders) | 104 | 95 | 85
Gfr (Metabolism and nutrition disorders) | 7 | 4 | 20
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 19 | 15 | 33
Alkalosis (Metabolism and nutrition disorders) | 0 | 1 | 2
Cholesterol,serum High (Metabolism and nutrition disorders) | 28 | 16 | 6
Proteinuria (Metabolism and nutrition disorders) | 62 | 65 | 60
Hemoglobinuria (Metabolism and nutrition disorders) | 1 | 2 | 3
Creatinine (Metabolism and nutrition disorders) | 43 | 33 | 132
Hypoalbuminemia (Metabolism and nutrition disorders) | 66 | 74 | 96
Gamma-Glutamyl Transferase (Ggt) (Metabolism and nutrition disorders) | 5 | 6 | 8
Alanine Aminotransferases (Alt) (Metabolism and nutrition disorders) | 98 | 109 | 77
Alkaline Phosphatase (Metabolism and nutrition disorders) | 61 | 86 | 73
Bilirubin (Metabolism and nutrition disorders) | 18 | 20 | 13
Lipase (Metabolism and nutrition disorders) | 0 | 1 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 14 | 9 | 22
Hypophosphatemia (Metabolism and nutrition disorders) | 44 | 32 | 38
Hyponatremia (Metabolism and nutrition disorders) | 97 | 113 | 141
Hyperuricemia (Metabolism and nutrition disorders) | 4 | 2 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 14 | 14 | 4
Creatine Phosphokinase (Cpk) (Metabolism and nutrition disorders) | 1 | 0 | 0
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 10 | 7 | 12
Amylase (Metabolism and nutrition disorders) | 1 | 1 | 5
Acidosis (Metabolism and nutrition disorders) | 3 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 15 | 13 | 9
Hypocalcemia (Metabolism and nutrition disorders) | 64 | 72 | 96
Hyperkalemia (Metabolism and nutrition disorders) | 28 | 28 | 49
Hyperglycemia (Metabolism and nutrition disorders) | 148 | 143 | 152
Hypokalemia (Metabolism and nutrition disorders) | 74 | 91 | 125
Hypoglycemia (Metabolism and nutrition disorders) | 30 | 28 | 31
Hypercalcemia (Metabolism and nutrition disorders) | 31 | 37 | 45
Hypomagnesemia (Metabolism and nutrition disorders) | 130 | 190 | 242
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 6 | 1
Fibrosis-Deep Connective Tissue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Seroma (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 6 | 15 | 12
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Device/Prosthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Joint-Function (Musculoskeletal and connective tissue disorders) | 19 | 23 | 15
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fracture (Musculoskeletal and connective tissue disorders) | 10 | 7 | 7
Fibrosis-Cosmesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Extremity-Upper (Function) (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Gait/Walking (Musculoskeletal and connective tissue disorders) | 8 | 9 | 4
Cervical Spine Rom (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 24 | 23 | 31
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 46 | 52 | 71
Muscle Weakness - Trunk (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Muscle Weakness - Right-Sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Muscle Weakness - Left-Sided (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Muscle Weakness - Extremity-Upper (Musculoskeletal and connective tissue disorders) | 6 | 12 | 11
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 20 | 30 | 17
Syncope (Nervous system disorders) | 5 | 12 | 24
Involuntary Movement (Nervous system disorders) | 15 | 25 | 10
Psychosis (Nervous system disorders) | 4 | 0 | 1
Myelitis (Nervous system disorders) | 0 | 0 | 1
Neurology - Other (Nervous system disorders) | 5 | 1 | 5
Mental Status (Nervous system disorders) | 0 | 2 | 4
Laryngeal Nerve Dysfunction (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 1 | 0
Cns Necrosis (Nervous system disorders) | 0 | 1 | 0
Mood Alteration - Euphoria (Nervous system disorders) | 0 | 2 | 0
Mood Alteration - Depression (Nervous system disorders) | 115 | 91 | 98
Mood Alteration - Anxiety (Nervous system disorders) | 111 | 102 | 122
Mood Alteration - Agitation (Nervous system disorders) | 8 | 11 | 6
Tremor (Nervous system disorders) | 12 | 13 | 21
Speech Impairment (Nervous system disorders) | 6 | 5 | 4
Seizure (Nervous system disorders) | 4 | 5 | 6
Personality (Nervous system disorders) | 2 | 1 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 2
Irritability (Nervous system disorders) | 2 | 1 | 2
Somnolence (Nervous system disorders) | 1 | 0 | 6
Cognitive Disturbance (Nervous system disorders) | 14 | 11 | 11
Cns Ischemia (Nervous system disorders) | 2 | 2 | 7
Ataxia (Nervous system disorders) | 5 | 8 | 4
Confusion (Nervous system disorders) | 18 | 10 | 15
Memory Impairment (Nervous system disorders) | 38 | 35 | 35
Dizziness (Nervous system disorders) | 113 | 107 | 111
Neuropathy,cranial - Cn Viii Hearing/Balance (Nervous system disorders) | 1 | 2 | 1
Neuropathy,cranial - Cn Vii Motor-Face (Nervous system disorders) | 0 | 1 | 0
Neuropathy,cranial - Cn V Motor-Jaw Muscles (Nervous system disorders) | 1 | 2 | 0
Neuropathy,cranial - Cn Ii Vision (Nervous system disorders) | 0 | 1 | 1
Neuropathy,cranial - Cn I Smell (Nervous system disorders) | 0 | 0 | 1
Neuropathy-Sensory (Nervous system disorders) | 406 | 394 | 407
Neuropathy-Motor (Nervous system disorders) | 48 | 56 | 35
Retinopathy (Eye disorders) | 1 | 0 | 0
Ocular/Visual - Other (Eye disorders) | 9 | 4 | 7
Vitreous Hemorrhage (Eye disorders) | 2 | 2 | 1
Nystagmus (Eye disorders) | 0 | 1 | 1
Nyctalopia (Eye disorders) | 2 | 0 | 0
Watery Eye (Eye disorders) | 26 | 26 | 8
Dry Eye (Eye disorders) | 16 | 18 | 12
Ocular Surface Disease (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 2 | 6 | 1
Photophobia (Eye disorders) | 4 | 3 | 3
Flashing Lights/Floaters (Eye disorders) | 18 | 23 | 17
Diplopia (Eye disorders) | 3 | 5 | 3
Blurred Vision (Eye disorders) | 89 | 82 | 78
Keratitis (Eye disorders) | 0 | 0 | 1
Eyelid Dysfunction (Eye disorders) | 3 | 2 | 4
Pain - Other (General disorders) | 18 | 41 | 31
Pain: Urethra (General disorders) | 14 | 29 | 14
Pain: Perineum (General disorders) | 2 | 4 | 1
Pain: Pelvis (General disorders) | 21 | 37 | 23
Pain: Breast (General disorders) | 2 | 4 | 5
Pain: Vagina (General disorders) | 12 | 9 | 12
Pain: Chest /Thorax Nos (General disorders) | 44 | 36 | 33
Pain: Chest Wall (General disorders) | 18 | 22 | 21
Pain: Throat/Pharynx/Larynx (General disorders) | 54 | 41 | 36
Pain: Pleura (General disorders) | 2 | 1 | 1
Pain: Larynx (General disorders) | 2 | 2 | 0
Pain: Eye (General disorders) | 6 | 5 | 4
Pain: Head/Headache (General disorders) | 234 | 201 | 209
Pain: Neck (General disorders) | 40 | 38 | 25
Pain: Intestine (General disorders) | 3 | 3 | 3
Pain: Extremity-Limb (General disorders) | 143 | 133 | 122
Pain: Buttock (General disorders) | 5 | 6 | 0
Pain: Back (General disorders) | 120 | 115 | 102
Pain: Joint (General disorders) | 235 | 210 | 199
Pain: Bone (General disorders) | 48 | 44 | 41
Pain: Lymph Node (General disorders) | 1 | 1 | 0
Pain: Gallbladder (General disorders) | 0 | 2 | 0
Pain: Kidney (General disorders) | 2 | 3 | 5
Pain: Bladder (General disorders) | 10 | 20 | 6
Pain: Pain Nos (General disorders) | 23 | 21 | 22
Pain: Stomach (General disorders) | 14 | 8 | 11
Pain: Rectum (General disorders) | 15 | 12 | 6
Pain: Peritoneum (General disorders) | 1 | 3 | 1
Pain: Oral Cavity (General disorders) | 28 | 23 | 14
Pain: Esophagus (General disorders) | 2 | 3 | 2
Pain: Dental/Teeth/Peridontal (General disorders) | 16 | 10 | 13
Pain: Abdominal Pain Nos (General disorders) | 243 | 311 | 346
Pain: Scalp (General disorders) | 5 | 3 | 6
Pain: Oral - Gums (General disorders) | 11 | 8 | 6
Pain: Skin (General disorders) | 6 | 7 | 4
Pain: Lip (General disorders) | 3 | 0 | 0
Pain: Middle Ear (General disorders) | 16 | 10 | 5
Pain: External Ear (General disorders) | 8 | 3 | 4
Pain: Cardiac/ Heart (General disorders) | 7 | 5 | 2
Pain: Face (General disorders) | 4 | 4 | 1
Pain: Muscle (General disorders) | 141 | 127 | 127
Pain: Anus (General disorders) | 4 | 6 | 1
Pain: Neuralgia (General disorders) | 11 | 10 | 6
Pain: Sinus (General disorders) | 9 | 10 | 4
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 6
Airway Obstruction - Trachea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Airway Obstruction - Bronchus (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 101 | 81 | 67
Edema, Larynx (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 11 | 7 | 5
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 75 | 57 | 58
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 3
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 143 | 147 | 116
Ards (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 7 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 202 | 203 | 143
Renal/Genitourinary - Other (Renal and urinary disorders) | 3 | 2 | 9
Stricture, Anastomotic, Gu - Ureter (Renal and urinary disorders) | 1 | 1 | 0
Prolapse Of Stoma, Gu (Renal and urinary disorders) | 0 | 1 | 0
Perforation, Gu - Vagina (Renal and urinary disorders) | 0 | 1 | 0
Leak, Gu - Vagina (Renal and urinary disorders) | 2 | 1 | 2
Leak, Gu - Bladder (Renal and urinary disorders) | 2 | 2 | 1
Cystitis (Renal and urinary disorders) | 10 | 15 | 7
Urinary Color Change (Renal and urinary disorders) | 3 | 3 | 0
Urinary Retention (Renal and urinary disorders) | 6 | 8 | 10
Urinary Electrolyte Wasting (Renal and urinary disorders) | 0 | 0 | 1
Obstruction, Gu - Ureter (Renal and urinary disorders) | 0 | 5 | 3
Obstruction, Gu - Bladder (Renal and urinary disorders) | 0 | 0 | 1
Incontinence, Urinary (Renal and urinary disorders) | 38 | 19 | 27
Fistula, Gu - Vagina (Renal and urinary disorders) | 1 | 2 | 0
Fistula, Gu - Genital Tract-Female (Renal and urinary disorders) | 0 | 0 | 1
Fistula, Gu - Bladder (Renal and urinary disorders) | 1 | 0 | 0
Bladder Spasm (Renal and urinary disorders) | 3 | 7 | 1
Renal Failure (Renal and urinary disorders) | 4 | 1 | 6
Urinary Frequency (Renal and urinary disorders) | 57 | 63 | 63
2nd Mal: Poss. Related To Cancer Rx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Libido (Reproductive system and breast disorders) | 12 | 5 | 4
Irregular Menses (Reproductive system and breast disorders) | 1 | 0 | 1
Vaginal Dryness (Reproductive system and breast disorders) | 24 | 10 | 19
Sexual/Reproductive Function: Other (Reproductive system and breast disorders) | 3 | 2 | 4
Vaginitis (Reproductive system and breast disorders) | 7 | 7 | 5
Vaginal Mucositis (Reproductive system and breast disorders) | 5 | 3 | 2
Vaginal Discharge (Reproductive system and breast disorders) | 21 | 19 | 22
Intra-Operative (Op) Injury: Nerves: Peripheral Motor Nos (Surgical and medical procedures) | 1 | 0 | 0
Intra-Op Injury: Teeth (Surgical and medical procedures) | 0 | 0 | 1
Intra-Op Injury: Nasal Cavity (Surgical and medical procedures) | 1 | 0 | 0
Intra-Op Injury: Kidney (Surgical and medical procedures) | 1 | 0 | 0
Intra-Op Injury: Small Bowel Nos (Surgical and medical procedures) | 0 | 1 | 0
Intra-Op Injury: Peritoneal Cavity (Surgical and medical procedures) | 0 | 1 | 0
Intra-Op Injury: Colon (Surgical and medical procedures) | 0 | 0 | 1
Intra-Op Injury: Abdomen Nos (Surgical and medical procedures) | 1 | 0 | 1
Intra-Op Injury: Adrenal Gland (Surgical and medical procedures) | 1 | 0 | 0
Syndromes - Other (General disorders) | 1 | 0 | 1
Cytokine Release Syndrome (General disorders) | 2 | 0 | 3
Flu-Like Syndrome (General disorders) | 12 | 9 | 12
Vascular - Other (Vascular disorders) | 1 | 0 | 1
Visceral Arterial Ischemia (Vascular disorders) | 1 | 0 | 0
Vein Injury - Other Nos (Vascular disorders) | 0 | 1 | 0
Peripheral Arterial Ischemia (Vascular disorders) | 0 | 0 | 1
Vein Injury - Extremity-Lower (Vascular disorders) | 1 | 0 | 0
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 7 | 5 | 10
Thrombosis/Thrombus/Embolism (Vascular disorders) | 21 | 27 | 30
Phlebitis (Vascular disorders) | 1 | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less